CLINICAL TRIAL: NCT00928824
Title: Dietary Nitrate in Japanese Traditional Foods Lowers Diastolic Blood Pressure in Healthy Volunteers.
Brief Title: Can Japanese Traditional Foods Lower Blood Pressure in Healthy Volunteers
Acronym: Horenso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Collaborators: Japanese Society for the Promotion of Science (Other)
Responsible Party: Prof Kamiya Shigeru, Kyorin Daigaku
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KyorinU
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: traditional Japanese diet — 10 days of nitrate rich diet (Japanese traditional). After that switch to nitrate low diet for 10 days (European foods). Study nitrate/nitrite in blood, saliva and blood pressure 3 times in each person (10 min each time). A list of Nitrate rich foods are provided.

SUMMARY:
The purpose of this study is to determine whether traditional japanese diet blood pressure in healthy volunteers.

DETAILED DESCRIPTION:
Japanese traditional diet contains considerably more nitrate/nitrite than the European foods. 80% of dietary nitrate originates from vegetables. Green leafy vegetables, especially spinach, salad and seaweed are rich in nitrates. Other vegetables contain nitrate at lower concentrations, but because they are consumed in greater quantity, they may contribute more nitrate and thus nitrite from the diet. Nitrate/nitrite is attributed multiple health benefits. Japanese people have an exceptional longevity and the lowest rate of heart diseases. On the other hand, gastric cancer rate is high too. Nitrate/nitrite is strongly correlated with these phenomena. Is this high nitrate consumption protective or damaging? Understanding dietary nitrite and nitrate consumption and its metabolism therefore becomes very important.

Aim: To compare conversion of nitrate to nitrite in Japanese people, measured in blood and in saliva during consumption of traditional Japanese foods vs European diet.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* high/low blood pressure

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin Univessity School of Medicine, Tokyo, Mitaka shi, Japan